CLINICAL TRIAL: NCT00659685
Title: Comparative, Randomized, Single-Dose, Cross Over Bioavailability of Kali's Ondansetron 16 mg ODT With That of GlaxoSmithKine's Zofran 16 mg ODT in Healthy, Male and Female Subjects Under Fasting Conditions
Brief Title: Bioavailability Study of Ondansetron 16 mg Orally Disintegrating Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Dr. Alfred Elvin/ Director Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ODO-P3-265
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: Bioequivalence; Ondansetron ODT; Fasting; To Determine Bioequivalence Under Fasting conditions
MeSH Terms: conditions — Fasting | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received Kali formulated products under fasting conditions
  Interventions: Drug: Ondansetron
- B (Active Comparator): Subjects received GlaxoSmithKline formulated products under fasting conditions
  Interventions: Drug: Zofran ODT

INTERVENTIONS:
Drug: Ondansetron — ODT, single-dose, fasting
  Other Names: Zofran ODT
  Arms: A
Drug: Zofran ODT
  Other Names: Ondansetron ODT
  Arms: B

SUMMARY:
Single-dose cross over comparative bioavailability of Ondansetron 16 mg ODT and Zofran 16 mg ODT

DETAILED DESCRIPTION:
To Compare the single-dose bioavailability of Kali's Ondansetron 16 mg ODT with that of GlaxoSmithKine's Zofran 16 mg ODT under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form(ICF) duly signed by the volunteer
* Males and females aged between 18 and 55 years with a body mass index (BMI) greater or equal to 19 and below 30 kg/ m2
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance(laboratory tests are presented in section 6.1.1.3)
* Healthy according to the laboratory results and physical examination.
* Non- or ex- smokers

Exclusion Criteria:

* Significant history of hypersensitivity to ondansetron or any related products as well as severe hypersensitivity reactions (like angioedema) to any drugs.
* Presence or history of significant gastrointestinal, liver or kidney disease, or any conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
* Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease.
* Females who are pregnant, lactating or are likely to become pregnant during the study phases.
* Females of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the body.
* Positive serum pregnancy test before and during the study.
* Maintenance therapy with any drug, or significant history or drug dependancy, alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic).
* Any clinically significant illness in the previous 28 days before day 1 of this study.
* Use of enzyme-modifying drugs in the previous 28 days before 1 day of this study (all barbiturates, corticosteroids, phenylhydantoins, etc.).
* Participation in another clinical trial in the previous 28 days before day 1 of this study.
* Donation of 500 mL of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study.
* Positive urine screening of drugs of abuse (drug names are presented in section 6.1.1.4).
* Positive results to HIV, HBsAg or anti-HCV tests.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-11

PRIMARY OUTCOMES:
Rate and Extend of absorption | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Christian Aumais, Principal Investigator — Algotithme Pharma Inc
Locations (1):
- Algorithme Pharma, Laval, Quebec, Canada